CLINICAL TRIAL: NCT06117527
Title: Placental Learning Model for Neurovascular Microsurgery for the Management of Intracranial Aneurysms
Acronym: NeuroVasc
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7907
Record Dates: First submitted 2022-11-14; First posted 2023-11-07 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Intracranial Aneurysm
Keywords: Intracranial aneurysm; Placental learning model; Neurovascular microsurgery; Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Training in microsurgical techniques for the management of intracranial aneurysms is carried out during the practical training of the DES in Neurosurgery and during the continuous training of neurosurgeons according to the indications of the patients of the department. Currently, the recent increase in indications for endovascular treatment compared to surgical indications has led to a decrease in surgical indications and in the experience of neurosurgeons. However, there are still surgical indications that are often complex situations that neurosurgeons must overcome with a specific simulation approach.

There are different simulation models for the treatment of intracranial aneurysms. The small animal (rodent) model has the disadvantage of being poorly suited to the reproduction of intracranial aneurysms (different extracranial vessel walls, too small intracerebral vessel caliber) and of being constraining to the establishment. The computerized stimulator model which has the advantage of being able to reproduce the anatomy of a patient but whose haptic sensitivity performance is difficult to reproduce for very fine movements, it is not very accessible because it is expensive. The placental model uses a fresh human placenta, the appearance of the vessels of which is very similar to those found intracerebrally, and dilations on their walls can be performed with a pediatric urinary catheter.

ELIGIBILITY:
Inclusion criteria:

* Woman over the age of 18;
* Placenta considered as surgical waste intended for incineration; with a negative infectious status verified during pregnancy follow-up
* Woman who did not express her opposition, after information, to the reuse of her placenta for educational purposes to improve the practical training of future neurosurgeons.

Exclusion criteria:

* Subject who expressed their opposition to participating in the study
* Subject under guardianship or curatorship
* Subject under safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Woman, over the age of 18, whose placenta from an adult woman, considered as surgical waste intended for incineration; with a negative infectious status verified during pregnancy follow-up
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-07-16 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the practical training of neurosurgery students | 1 month after training students in microsurgery for brain aneurysms
  Hands-on training will be assessed by the Brain Aneurysm Microsurgery Skills Rating Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Neurochirurgie - CHU de Strasbourg - France, Strasbourg, France